CLINICAL TRIAL: NCT04520347
Title: An International VT Ablation Center Collaborative Group (IVTCC): A Multicenter Ventricular Tachycardia Catheter Ablation Registry
Brief Title: IVTCC 2.0: A Prospective Multicenter Ventricular Tachycardia Catheter Ablation Registry
Acronym: IVTCC
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jason Bradfield, MD, Director, Specialized Program for Ventricular Tachycardia, University of California, Los Angeles
Other Study IDs: 17-001725
Record Dates: First submitted 2020-07-10; First posted 2020-08-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Ventricular Arrhythmia; Ventricular Tachycardia; Premature Ventricular Contraction (PVC); Cardiomyopathy
Keywords: Arrhythmia; Cardiac Conduction System Disease; Sudden Cardiac Death; Implantable Cardiac Defibrillator (ICD)
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Premature Complexes; Cardiomyopathies; Arrhythmias, Cardiac; Cardiac Conduction System Disease; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective multi-center international registry. The objective of this registry is to collect prospective data on patients undergoing catheter ablation for Ventricular Tachycardia (VT) and Premature Ventricular Contractions (PVC). The registry will be used for clinical monitoring, research, and quality improvement purposes.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD), predominantly due to ventricular tachyarrhythmias, is a leading cause of mortality in the United States and around the world. Catheter ablation of ventricular arrhythmias has proven efficacious in reducing the burden of arrhythmias and reducing implantable cardiac defibrillator (ICD) shocks.

The aim of this study is to create a prospective international database registry that will allow for better assessment of the outcomes of catheter ablation of ventricular arrhythmias. The registry, with approximately 30 participating centers, will help to identify the overall success rates and associated benefits of the procedure and provide more comprehensive data on understudied populations and treatment.

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing catheter ablation for ventricular tachycardia (VT) or premature ventricular contractions (PVCs).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ventricular arrhythmias that undergo catheter ablation for ventricular tachycardia or premature ventricular contractions.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Ventricular tachycardia (VT) recurrence | From date of procedure assessed by shock, Anti-Tachycardia Pacing, or repeat procedure, up to 10 years.
  Freedom from ventricular tachycardia episodes requiring ICD Intervention (shock or Anti-Tachycardia Pacing) or repeat procedure.

SECONDARY OUTCOMES:
Rate of complications | From date of procedure assessed up to 12 months.
  Cardiovascular-related and procedure-related major complications and/or adverse events.
Time to transplant or death | From date of procedure assessed by date of transplant and/or death, up to 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Bradfield, MD, Principal Investigator — University of California, Los Angeles; Kalyanam Shivkumar, MD, PhD, Study Chair — University of California, Los Angeles; Paolo Della Bella, MD, Study Chair — San Raffaele Hospital, Italy; Francis Marchlinski, MD, FACC, FAHA, FHRS, Study Chair — University of Pennsylvania Health System; Andrea Natale, MD, FACC, FHRS, FESC, Study Chair — Texas Cardiac Arrhythmia Institute at St. David's Medical Center; William G Stevenson, MD, Study Chair — Vanderbilt Heart and Vascular Institute
Locations (41):
- United States (34):
  - Banner Health, University of Arizona Medical Center, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford HealthCare, Hartford, Connecticut
  - University of Florida Health, Gainesville, Florida
  - The Kansas City Heart Rhythm Institute, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Heart and Vascular Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Health Care, Worcester, Massachusetts
  - University of Michigan Frankel Cardiovascular Center, Ann Arbor, Michigan
  - University of Minnesota VA Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - The Mount Sinai Hospital, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Wellspan Health, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Institute at St. David's Medical Center, Austin, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
- The Montreal Heart Institute, Montreal, Canada
- Shaare Zedek Medical Center, Jerusalem, Israel
- Dokkyo Medical University Koshigaya Hospital, Koshigaya, Japan
- Netherlands (2):
  - Leiden University, Leiden
  - Erasmus Medical Center, Rotterdam
- Gregorio Marañón General University Hospital, Madrid, Spain
- St. George's Hospital, Wandsworth, United Kingdom